CLINICAL TRIAL: NCT00444938
Title: Evaluation of the H-Coil (TMS) Device - Safety and Feasibility in Bipolar Depression
Brief Title: Evaluation of the H-Coil Transcranial Magnetic Stimulation (TMS) Device in the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH-50506
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2007-03

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: H1 -coil TMS device

SUMMARY:
This study is evaluating the potential antidepressive effect of a 4 week treatment protocol using the H-coil deep TMS device in bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar depression

Exclusion Criteria:

* No other axis I disorder
* Risk factors for convulsions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiran V Harel, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel

REFERENCES:
- [Derived] Harel EV, Zangen A, Roth Y, Reti I, Braw Y, Levkovitz Y. H-coil repetitive transcranial magnetic stimulation for the treatment of bipolar depression: an add-on, safety and feasibility study. World J Biol Psychiatry. 2011 Mar;12(2):119-26. doi: 10.3109/15622975.2010.510893. Epub 2010 Sep 21. PMID 20854181